CLINICAL TRIAL: NCT07391449
Title: Heart Rate Variability Guided Optimization of Physical Activity and Exercise Prescription to Enhance Rehabilitation Outcomes in Individuals With Knee Osteoarthritis (HOPE-OA Trial)
Brief Title: Heart Rate Variability Guided Physical Activity and Exercise Prescription in Individuals With Knee Osteoarthritis
Acronym: HOPE-OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shahnawaz Anwer, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20251219004
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; HRV; Physical activity; Home exercise; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV guided home exercise (Experimental)
  Interventions: Behavioral: HRV-guided home exercise prescription
- Traditional home exercise (Active Comparator)
  Interventions: Behavioral: Traditional Home Exercise

INTERVENTIONS:
Behavioral: HRV-guided home exercise prescription — Participants in this group will follow the same exercise structure as the traditional home exercise group; however, their exercise program will be individualised according to daily HRV profiles. Exercise sessions will be performed three times per week for 12 weeks (36 sessions). All participants will conduct HRV measurements, starting one week before the intervention and continuing until its completion. HRV will be measured each morning immediately after awakening and bladder voiding, with participants remaining in the supine position for 5 minutes. The validated smartphone application, "HRV4Training" (http://www.hrv4training.com/) will be used to record HRV data [31]. The analysis provides the root mean square of successive differences between R-R intervals (root mean square successive differences [rMSSD]), derived via photoplethysmography. A 7-day rolling average (Ln rMSSD7d) will be computed, and HRV parameters will be calculated.
  Arms: HRV guided home exercise
Behavioral: Traditional Home Exercise — Participants in this group will measure their HRV daily as described in the next section; however, these HRV measurements will not be used to guide their exercise prescription. Instead, participants will follow a standardized home exercise programme, conducted three sessions per week for 12 weeks (36 sessions). Each session will include a 5-10-minute warm-up, a main exercise component comprising aerobic, strengthening, and stretching exercises (e.g., stretching of lower extremity muscles including knee extensors, knee flexors, and calf), and a 5-minute cooldown [27-29]. The warm-up phase will comprise mobility exercises designed to activate the lower extremity muscles, particularly the quadriceps and hamstrings, while the cool-down will incorporate stretching the muscle groups engaged during the session.
  Arms: Traditional home exercise

SUMMARY:
The aim of this trial is to conduct a 12-week randomised controlled trial comparing an HRV-guided home exercise program with traditional home exercise program for individuals with knee osteoarthritis (KOA), followed by 24-week assessment. The trial employs a validated HRV sensor and the HRV4Training app to record daily HRV measurements, enabling personalized exercise intensity adjustments. Participants with high HRV are prescribed high-intensity exercises, while those with low HRV undertake low-intensity exercises. In contrast, the traditional exercise group follows a standardised program, progressing from low to high intensity over the 12-week period.

The primary objective of this trial is to evaluate the effect of HRV-guided exercise on pain and functional disability in patients with KOA using validated outcome measures assessed at baseline, 12 weeks (post-intervention), and 24 weeks. Longitudinal semi-structured qualitative interviews at weeks 12 and 24 will explore participants' experiences and perceived barriers to exercise adherence. A mediation analysis will elucidate the physiological mechanisms underlying the efficacy of HRV-guided exercise. Secondary objectives include comparing HRV-guided and traditional home exercise programme in terms of exercise adherence, quality of life, sleep quality, self-efficacy, patient satisfaction, physical performance, balance, muscle strength, and lower limb biomechanics. Exploratory aims involve evaluating long-term effects (up to 24 weeks), examining associations between baseline HRV profiles and key outcomes, and determining the cost-effectiveness of HRV-guided exercise relative to traditional programme. The trial employs a robust methodological design, applying mixed-effects models and an intention-to-treat approach for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will include adults aged 45 years and older with symptomatic KOA, diagnosed according to the American College of Rheumatology Clinical Criteria for the Classification and Reporting of KOA.
2. Mild to moderate KOA (Kellgren Lawrence grade ≤ grade III),
3. a body mass index (BMI) ≤ 40 kg/m2, and
4. an average knee pain intensity ≥ 3 on a 0-10 numerical rating scale during the past week.

Exclusion Criteria:

1. presence of neurological disorders;
2. nonambulatory status;
3. implanted electrical devices;
4. systemic inflammatory arthritis (e.g., gout);
5. significant cognitive impairment;
6. prior hip or knee arthroplasty;
7. history of trauma or surgical arthroscopy of either knee within the past six months;
8. participation in a similar study within the past six months;
9. engagement in an exercise programme within the past six months;
10. receipt of knee intra-articular injection within the past three months;
11. current anticoagulant therapy;
12. recent or planned surgery within three months; and
13. any medical comorbidities precluding safe participation in exercise.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee pain | change from pre- to post-treatment (12 weeks)
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale. Higher scores mean more discomfort. The WOMAC pain subscale include five items for pain (scores range from 0 to 20).
Physical Function | Change from pre- to post-treatment (12 weeks)
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale. Higher scores mean more difficulty with daily tasks. The WOMAC function subscale include 17 items for functional restriction (scores range from 0 to 68).

SECONDARY OUTCOMES:
Healthcare resource utilisation | week 12 and week 24
  Client service recipient inventory (CSRI) will utilised to assess healthcare resource utilisation.
Quality adjusted life year (QALY) | week 12 and week 24
  Quality-adjusted life-years (QALYs) will serve as outcome metric for economic evaluation, derived from the 5-level EuroQol instrument (EQ-5D-5L). Unadjusted mean costs and cost differences between HRV-G and TRD-G exercise groups will be examined for aggregate and disaggregated cost components, including intervention costs, healthcare service use, and pharmaceutical expenditures. Total cost differences (ΔC) and effect differences (ΔE) will be estimated, adjusting for baseline demographic and health characteristics. Responses from the EQ-5D-5L will be converted into utility scores, which will then be used to calculate QALY changes over the study period. The incremental cost-effectiveness ratio (ICER) will be computed using the formula ICER = ΔC/ΔE.
Knee pain | changes from baseline to week 24
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale. Higher scores mean more discomfort. The WOMAC pain subscale include five items for pain (scores range from 0 to 20).
Physical function | changes from baseline to week 24
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale. Higher scores mean more difficulty with daily tasks. The WOMAC function subscale include 17 items for functional restriction (scores range from 0 to 68).
Arthritis self-efficacy scale (ASES) | Baseline, week 12, week 24
  The Arthritis self-efficacy scale (ASES) consists of 20 items that assess a patient's confidence in controlling pain, physical function, and other disease-related factors. The scale has three parts: pain management, function, and other symptoms like fatigue. Each question asks the respondent to rate their self-efficacy on a scale from 10 to 100, with 10 meaning "very uncertain" and 100 meaning "very certain" about their capacity to do particular tasks or deal with symptoms. Therapists give the questionnaire to patients and tell them to think about how confident they usually feel during the past week when they answer. To get subscale scores, the scores in each domain are added together. Higher scores indicate greater perceived self-efficacy.
Pittsburgh Sleep Quality Index | Baseline, week 12, week 24
  The Pittsburgh Sleep Quality Index (PSQI) used to measure the quality and patterns of sleep in adults. It identify sleep quality between "poor" and "good" sleep by utilizing seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. A lower PSQI score indicates better sleep quality, with scores of ≤5 considered good and ≥5 indicating poor sleep quality.
Center for Epidemiologic Studies Depression Scale (CESD) | Baseline, week 12, week 24
  The Center for Epidemiologic Studies Depression Scale (CESD) is a widely used self-report scale designed to measure depressive symptoms in the general population, consisting of 20 items that assess how often individuals have experienced specific symptoms over the past week. The score is the sum of the 20 questions. Possible range is 0-60. A score of 16 points or more is considered depressed.
Patient Specific Functional Scale (PSFS) | Baseline, week 12, week 24
  The Patient Specific Functional Scale (PSFS) is a self-reported valid, reliable, and responsive outcome measure for patients with back, neck, knee and upper extremity problems. It has also been shown to have a high test-retest reliability in both generic lower back pain and knee dysfunction issues. It is also clinically responsive to changes over time with chronic pain patients. Patients are asked to identify up to five important activities they are unable to perform or are having difficulty with as a result of their problem eg putting socks on, shopping. Patients are asked to rate their current level of difficulty associated with each activity on an 11-point scale from 0 (unable to perform) to 10 (able to perform at prior level). Higher the score better the function.
30 second chair stand test (30sCST) | changes from baseline to week 12
  The 30 second chair stand test (30sCST) requires participants to rise fully from a seated position in an unarmed, straight-backed chair (seat height: 45 cm) and return to a seated position until fully seated. The total number of chair-stand repetitions performed within a 30-s interval will be recorded. Participants will engage in two slow-paced practice repetitions prior to formal testing to ensure comprehension.
40-m fast-paced walk test (40MFPW) | changes from baseline to week 12
  The 40-m fast-paced walk test (40MFPW) requires participants to walk as quickly and safely as possible along a 10-m walkway, turning around a cone positioned 2 m beyond each end of the walkway, resulting in a total distance of 40 m. Participants may utilize a walking aid if necessary, and the duration for task completion will be documented [22].
Stair-climbing test (SCT) | changes from baseline to week 12
  The stair-climbing test (SCT) will require participants to ascend and descend nine stairs, each with a step height of 20 cm, as quickly as possible while ensuring safety. A handrail will be provided for participants who wish to utilize it or require walking aids. The duration for participants to complete the ascending and descending tasks will be recorded.
Gait analysis | changes from baseline to week 12
  Motion capture system will be utilized for gait assessment.
Quadriceps and Hamstring muscle strength | changes from baseline to week 12
  An isokinetic dynamometry will be used for the assessment of Quadriceps and Hamstring muscle strength
Single and double leg standing balance | changes from baseline to week 12
  Bertec balance system will be used for the assessment of Single and double leg standing balance.
Heart rate variability (HRV) | Daily
  All participants will conduct HRV measurements, starting one week before the intervention and continuing until its completion. HRV will be measured each morning immediately after awakening and bladder voiding, with participants remaining in the supine position for 5 minutes. The validated smartphone application, "HRV4Training" (http://www.hrv4training.com/) will be used to record HRV data [31]. The analysis provides the root mean square of successive differences between R-R intervals (root mean square successive differences [rMSSD]), derived via photoplethysmography. The rMSSD is preferred for its reliability over other HRV indices. To normalise data distribution, HRV values will be log-transformed using the natural logarithm (Ln) before statistical analysis. A 7-day rolling average (Ln rMSSD7d) will be computed, and HRV parameters will be calculated during both the familiarization period and on a weekly basis throughout the experimental phase.

OTHER OUTCOMES:
System Usability Scale (SUS) | week 12
  The feasibility and usability of the HRV device for optimising home exercise programme will be evaluated using the System Usability Scale (SUS). The HRV device will be considered a viable tool for rehabilitation and home exercise optimization in individuals with KOA if it achieves an average SUS score of 70 points or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Shanawaz Anwer, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Department of Rehabilitation Sciences, The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data that underlie the results reported in publication(s).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following publication(s).
Access Criteria: Data will only be available for individual participant data. Data will be disseminated to researchers who submit a methodologically rigorous proposal and whose intended usage of the data has received approval from an independent review committee designated for this purpose.

REFERENCES:
- [Background] 37. Saldaña J. Longitudinal qualitative research: analyzing change through time. Bloomsbury Publishing PLC; 2003 May 16.
- [Background] 36. Plano Clark VL, Schumacher K, West C, Edrington J, Dunn LB, Harzstark A, Melisko M, Rabow MW, Swift PS, Miaskowski C. Practices for embedding an interpretive qualitative approach within a randomized clinical trial. Journal of Mixed Methods Research. 2013 Jul;7(3):219-42.
- [Background] 35. Winser SJ, Pang M, Whitney S, Chan AY, Chen C. Cost and effectiveness of Dual-task training on balance and fall risk in individuals with cerebellar ataxia: A randomized controlled trial. Physiotherapy. 2024 Jun 1;123:e113.
- [Background] 34. LaFlair GT, Egbert J, Plonsky L. A practical guide to bootstrapping descriptive statistics, correlations, t tests, and ANOVAs. Advancing quantitative methods in second language research. 2015 Jul 3;46.
- [Background] 33. Lewis JR. The system usability scale: past, present, and future. International Journal of Human-Computer Interaction. 2018 Jul 3;34(7):577-90.
- [Background] 32. Vesterinen V, Häkkinen K, Laine T, Hynynen E, Mikkola J, Nummela A. Predictors of individual adaptation to high-volume or high-intensity endurance training in recreational endurance runners. Scandinavian journal of medicine & science in sports. 2016 Aug;26(8):885-93.
- [Background] 31. Plews DJ, Scott B, Altini M, Wood M, Kilding AE, Laursen PB. Comparison of heart-rate-variability recording with smartphone photoplethysmography, polar H7 chest strap, and electrocardiography. International journal of sports physiology and performance. 2017 Nov 1;12(10):1324-8.
- [Background] 30. Williams N. The Borg rating of perceived exertion (RPE) scale. Occupational medicine. 2017 Jul 1;67(5):404-5.
- [Background] 29. Alghadir AH, Anwer S, Sarkar B, Paul AK, Anwar D. Effect of 6-week retro or forward walking program on pain, functional disability, quadriceps muscle strength, and performance in individuals with knee osteoarthritis: a randomized controlled trial (retro-walking trial). BMC musculoskeletal disorders. 2019 Apr 9;20(1):159.
- [Background] 28. Anwer S, Alghadir A, Brismee JM. Effect of home exercise program in patients with knee osteoarthritis: a systematic review and meta-analysis. Journal of geriatric physical therapy. 2016 Jan 1;39(1):38-48.
- [Background] 27. Anwer S, Alghadir A. Effect of isometric quadriceps exercise on muscle strength, pain, and function in patients with knee osteoarthritis: a randomized controlled study. Journal of physical therapy science. 2014;26(5):745-8.
- [Background] 26. Fritz MS, MacKinnon DP. Required sample size to detect the mediated effect. Psychological science. 2007 Mar;18(3):233-9. 27. Anwer S, Alghadir A. Effect of isometric quadriceps exercise on muscle strength, pain, and function in patients with knee osteoarthritis: a randomized controlled study. Journal of physical therapy science. 2014;26(5):745-8.
- [Background] 25. Rizvi MR, Sharma A, Hasan S, Ahmad F, Asad MR, Iqbal A, Alghadir AH. Exploring the impact of integrated polyvagal exercises and knee reinforcement in females with grade II knee osteoarthritis: a randomized controlled trial. Scientific Reports. 2023 Nov 3;13(1):18964.
- [Background] 24. Williams A, van Dongen JM, Kamper SJ, O'Brien KM, Wolfenden L, Yoong SL, Hodder RK, Lee H, Robson EK, Haskins R, Rissel C. Economic evaluation of a healthy lifestyle intervention for chronic low back pain: A randomized controlled trial. European Journal of Pain. 2019 Mar;23(3):621-34.
- [Background] 23. Jackson D, McCrone P, Mosweu I, Siegert R, Turner-Stokes L. Service use and costs for people with long-term neurological conditions in the first year following discharge from in-patient neuro-rehabilitation: a longitudinal cohort study. PLoS One. 2014 Nov 17;9(11):e113056.
- [Background] 22. Joudeh AA, Alghadir AH, Zafar H, Elwatidy SM, Tse C, Anwer S. Effect of quadriceps and calf muscles fatigue on standing balance in healthy young adult males. Journal of Musculoskeletal & Neuronal Interactions. 2018 Jun;18(2):248.
- [Background] 21. Sun J, Liu Y, Yan S, Cao G, Wang S, Lester DK, Zhang K. Clinical gait evaluation of patients with knee osteoarthritis. Gait & posture. 2017 Oct 1;58:319-24.
- [Background] 20. Dobson F, Bennell KL, Hinman RS, Abbott JH, Roos EM. Recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. OARSI 2013. https://oarsi.org/sites/oarsi/files/docs/2013/manual.pdf. Accessed 2 October 2025.
- [Background] 19. Stratford P, Gill C, Westaway M, Binkley J. Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy Canada. 1995 Oct;47(4):258-63.
- [Background] 17. Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Quality of Life Research. 2005 Oct;14(8):1943-52.
- [Background] 16. Brand E, Nyland J, Henzman C, Mcginnis M. Arthritis self-efficacy scale scores in knee osteoarthritis: a systematic review and meta-analysis comparing arthritis self-management education with or without exercise. Journal of Orthopaedic & Sports Physical Therapy. 2013 Dec;43(12):895-910.
- [Background] 15. Myers BJ. Isokinetic testing of muscle strength in older adults with knee osteoarthritis: an integrative review. Isokinetics and Exercise Science. 2020 Aug;28(3):269-90.
- [Background] 14. Marriott KA, Hall M, Maciukiewicz JM, Almaw RD, Wiebenga EG, Ivanochko NK, Rinaldi D, Tung EV, Bennell KL, Maly MR. Are the effects of resistance exercise on pain and function in knee and hip osteoarthritis dependent on exercise volume, duration, and adherence? A systematic review and meta-analysis. Arthritis Care & Research. 2024 Jun;76(6):821-30.
- [Background] 13. Rodrigues JA, Santos BC, Medeiros LH, Gonçalves TC, Júnior CR. Effects of different periodization strategies of combined aerobic and strength training on heart rate variability in older women. The Journal of Strength & Conditioning Research. 2021 Jul 1;35(7):2033-9.
- [Background] 12. Symonds T, Hughes B, Liao S, Ang Q, Bellamy N. Validation of the Chinese Western Ontario and McMaster universities osteoarthritis index in patients from mainland China with osteoarthritis of the knee. Arthritis care & research. 2015 Nov;67(11):1553-60.
- [Background] 11. Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. Bmj. 2014 Mar 7;348.
- [Background] 10. Chan AW, Tetzlaff JM, Gøtzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hróbjartsson A, Schulz KF, Parulekar WR, Krleža-Jerić K. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. Bmj. 2013 Jan 9;346.
- [Background] 9. Morinaga H, Takai Y. Heart rate variability-guided aerobic training without moderate-intensity enhances submaximal and maximal aerobic power with less training load. Journal of Human Sport and Exercise. 2025;20(1):366-80.
- [Background] 8. Düking P, Zinner C, Trabelsi K, Reed JL, Holmberg HC, Kunz P, Sperlich B. Monitoring and adapting endurance training on the basis of heart rate variability monitored by wearable technologies: A systematic review with meta-analysis. Journal of Science and Medicine in Sport. 2021 Nov 1;24(11):1180-92.
- [Background] 7. Carrasco-Poyatos M, Granero-Gallegos A, López-García GD, López-Osca R. HRV-guided training for elders after stroke: a protocol for a cluster-randomized controlled trial. International journal of environmental research and public health. 2022 Aug 31;19(17):10868.
- [Background] 6. Ortigosa-Márquez JM, Reigal RE, Portell M, Morales-Sánchez V, Hernández-Mendo A. Observación automatizada: La variabilidad de la frecuencia cardíaca y su relación con las variables psicológicas determinantes del rendimiento en nadadores jóvenes. Anales de Psicología/Annals of Psychology. 2017 Jul 21;33(3):436-41.
- [Background] 5. Hawker GA. Osteoarthritis is a serious disease. Clin Exp Rheumatol. 2019 Sep 1;37(Suppl 120):3-6.
- [Background] 4. The Chinese University of Hong Kong. Osteoarthritis in Hong Kong Chinese-prevalence, aetiology and prevention. 2001. Available from: http://www.cuhk.edu.hk/ipro/010306e.htm. Accessed 07 Oct 2025.
- [Background] 3. Liu Q, Wang S, Lin J, Zhang Y. The burden for knee osteoarthritis among Chinese elderly: estimates from a nationally representative study. Osteoarthritis and cartilage. 2018 Dec 1;26(12):1636-42.
- [Background] 2. Steinmetz JD, Culbreth GT, Haile LM, Rafferty Q, Lo J, Fukutaki KG, Cruz JA, Smith AE, Vollset SE, Brooks PM, Cross M. Global, regional, and national burden of osteoarthritis, 1990-2020 and projections to 2050: a systematic analysis for the Global Burden of Disease Study 2021. The Lancet Rheumatology. 2023 Sep 1;5(9):e508-22.
- [Background] 1. Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. British journal of sports medicine. 2015 Dec 1;49(24):1554-7.